CLINICAL TRIAL: NCT03579069
Title: Does the Performance of the Ductus Venosus Doppler at 16 Weeks Allow to Increase the Screening of the Twin-twin Transfusion Syndrome and to Reduce the Neonatal Mortality?
Brief Title: Ductus Venosus Doppler at 16 Weeks in Monochorial Pregnancy
Acronym: DVSTT
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0254
Record Dates: First submitted 2018-06-12; First posted 2018-07-06 (Actual); Last update posted 2019-04-18 (Actual); Status verified 2018-06

CONDITIONS: Twin Pregnancy, Monochorionic; Pregnancy Followed
Keywords: Ductus venosus Doppler

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Ductus venosus Doppler realized: Ductus venosus Doppler realized
  Interventions: Other: Ductus venosus Doppler
- Ductus venosus Doppler unrealized: Ductus venosus Doppler unrealized

INTERVENTIONS:
Other: Ductus venosus Doppler — Ductus venosus Doppler
  Groups: Ductus venosus Doppler realized

SUMMARY:
Studies shows that the realization of the Ductus venosus Doppler may improve the screening of the twin-twin transfusion syndrome. In this study, we want to compare the outcome of monochorial pregnancy when this Doppler was performed during the ultrasound at16 weeks, and when it wasn't. In order to do that, we will compile past reports (January 2015/ January 2018) of all monochorial pregnancy handled in the hospital of Montpellier and Kremlin Bicêtre. We will establish if the Doppler was done or not, if the twin-twin transfusion syndrome appears and the neonatal outcome.

ELIGIBILITY:
Inclusion criteria:

* Monochorionic diamniotic twin pregnancies
* Monochorionicity diagnosed at the first-trimester
* Follow up and ultrasound realized at the hospital of Montpellier or Kremlin Bicêtre
* Screening for twin-twin transfusion syndrome achieved

Exclusion criteria:

* Missing ultrasound
* Unregistered outcome of the pregnancy
* Eclampsia and pre-eclampsia

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Monochorial pregnancy followed in the hospital of Montpellier or Bicêtre
Sampling Method: Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2018-07-30 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Occurrence of a twin to twin transfusion syndrome | 1 day
  Occurrence of a twin to twin transfusion syndrome during pregnancy

SECONDARY OUTCOMES:
neonatal mortality rate | 1 day
  neonatal mortality rate

CONTACTS AND LOCATIONS:
Overall Officials: Celine FOREL, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uhmontpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC